CLINICAL TRIAL: NCT03033979
Title: Prolonged Use of the Laryngeal Mask Airway ProSealTM: a Report of Seven Cases Lasting 5-11 Hours
Brief Title: Prolonged Laryngeal Mask Airway ProSealTM Use
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Other Study IDs: Schulthess_Anä_9
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Airway Management

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators conclude that use of the LMA ProSealTM for prolonged procedures is feasible. In principle, it should be safer and more effective than the LMA ClassicTM provided basic guidelines are followed.

DETAILED DESCRIPTION:
There is controversy concerning use of the classic laryngeal mask airway (LMA ClassicTM) for prolonged procedures, particularly over 2 hours, as some clinicians consider it unsuitable for positive pressure ventilation (needed to counter the alleged progressive respiratory fatigue with time) and/or unsuitable for airway protection (needed to counter the alleged progressive increase in aspiration risk with time). The LMA ProSealTM is a laryngeal mask device with a modified cuff to facilitate ventilation and a drain tube to provide airway protection. In principle, the LMA ProSealTM should be more suitable than the LMA ClassicTM for prolonged procedures; however, there are only four reports and one case series.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 - 3
* Age 19-85 yr
* Written informed consent

Exclusion Criteria:

* Difficult airway
* Non fasted
* BMI > 35

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We describe the use of the LMA ProSealTM in seven patients in a variety of clinical situations for procedures lasting more than 5 hours.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the LMA ProSealTM for prolonged use | 30 Minutes
  Oropharyngeal leak pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Christian Keller MD, M.Sc., Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No